CLINICAL TRIAL: NCT00851786
Title: A Phase II, Randomized, Double-Blind, Placebo-Controlled Clinical Trial to Evaluate the Safety, Tolerability, and Immunogenicity of ZOSTAVAX® (Zoster Vaccine Live) in Human Immunodeficiency Virus (HIV)-1-Infected Adults on Potent Combination ART With Conserved Immune Function
Brief Title: Live Zoster Vaccine in HIV-Infected Adults on Antiretroviral Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Adult AIDS Clinical Trials Group (Network); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: A5247; 10519 (Registry Identifier: DAIDS ES Registry ID); ACTG A5247
Record Dates: First submitted 2009-02-25; First posted 2009-02-26 (Estimated); Results first posted 2012-10-10 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2018-01

CONDITIONS: Herpes Zoster; HIV Infections
Keywords: Herpes Zoster Vaccine; Herpes Zoster Virus; HIV
MeSH Terms: conditions — Herpes Zoster; HIV Infections; Chickenpox | interventions — Herpes Zoster Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Participants with CD4 cell counts of 200 cells/uL or greater in Stages 1 and 2, stratified by CD4 cell counts (200-349 cells/uL vs. >=350 cells/uL), will be given one dose of ZOSTAVAX (Zoster Vaccine Live) at Day 0 and Week 6 and will be followed for at least 42 days after each vaccination after which a safety assessment will be conducted.
  Interventions: Biological: ZOSTAVAX
- 2 (Placebo Comparator): Participants with CD4 cell counts of 200 cells/uL or greater in Stages 1 and 2, stratified by CD4 cell counts (200-349 cells/uL vs. >=350 cells/uL), will be given one dose of placebo at Day 0 and Week 6 and will be followed for at least 42 days after each vaccination after which a safety assessment will be conducted
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: ZOSTAVAX — Subcutaneous injection of 0.65 mL of ZOSTAVAX at Day 0 and Week 6
  Arms: 1
Biological: Placebo — Subcutaneous injection of 0.65 mL of placebo at Day 0 and Week 6
  Arms: 2

SUMMARY:
Herpes zoster, or shingles, is the result of a viral infection that causes a painful skin rash, usually in older people or people with suppressed immune systems like those infected with HIV. The ZOSTAVAX vaccine has been shown to reduce the number of infections and symptoms of herpes zoster infection in people over the age of 60. The purpose of this study is to evaluate the safety, tolerability, and immunogenicity of two doses of ZOSTAVAX in HIV-1-infected adults with conserved immune function (Cd4+ T cell counts >=200 cells/uL) virologically suppressed on potent combination antiretroviral therapy (ART).

DETAILED DESCRIPTION:
The varicella-zoster virus (VZV) which causes herpes zoster (HZ), or shingles, is associated with a painful skin rash and post-herpetic neuralgia (PHN). The incidence and severity of HZ and PHN increase as immune function decreases, as in elderly or HIV-infected people. The live VZV vaccine, ZOSTAVAX, has been shown to reduce the incidence and severity of HZ and PHN in people over the age of 60. The main purpose of this study is to determine whether a two-dose regimen of ZOSTAVAX is safe and well-tolerated in HIV-infected individuals with conserved immune function.

This study has two stages and two arms. It may last up to 24 weeks per subject. In Stage 1, 48 participants with CD4 cell counts of 200 or more cells/uL will be enrolled (24 participants with a CD4 count between 200 and 349 cells/uL and 24 participants with a CD4 count equaling 350 or more cells/uL). These participants will be randomized 3:1 to receive two doses of ZOSTAVAX or placebo at least six weeks apart. If certain safety criteria are met for Stage 1, enrollment will be opened to Stage 2. Stage 2 will enroll approximately 352 subjects with CD4+ T cell counts >= 200 cells/uL. In Stage 2, participants will be stratified using the same parameters as Stage 1 and will then be randomized 3:1 to receive either two doses of vaccine or placebo according to the same schedule. Participants will be followed for at least 42 days after each vaccination. Temperatures will be collected daily for 42 days following each vaccination. Telephone contact will also be made 2 to 3 days after each vaccination and at 24 weeks following the initial vaccination to obtain information regarding vaccination-related symptoms.

All participants will have between 6 and 8 study visits. At the screening visit, documentation of HIV status is required, and blood and urine collection, a physical exam, medical history, and clinical assessment will occur. At each visit, a targeted physical exam will occur. At some visits, blood and urine collection, and a clinical assessment will occur. Antiretroviral medications are not provided by this study.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected
* Use of potent combination ART regimen within 90 days prior to entry and undetectable plasma HIV RNA level within 90-210 days prior to study entry
* CD4 cell count of at least 200 cells/uL obtained within 30 days prior to study entry
* Laboratory values obtained within 90 days prior to study entry

  * Hemoglobin 7.0 g/dL or greater
  * Platelet count 50,000/mm3 or greater
  * Creatinine 3 x ULN or less
  * AST (SGOT), ALT (SGPT), and alkaline phosphatase 5 x ULN or less
* For females of reproductive potential, a negative serum or urine pregnancy test within 24 hours prior to study entry
* Willing to use accepted forms of contraception for the duration of the study
* History of varicella or herpes zoster more than 1 year prior to vaccination or VZV seropositivity at any time prior to entry
* Men and women age >=18 years
* Ability and willingness of subject or legal guardian/representative to provide informed consent

Exclusion Criteria:

* History of nadir CD4+ count <100 cells/uL
* Known or suspected immune dysfunction caused by a medical condition or any cause other than HIV infection, such as congenital immunodeficiency, organ or bone marrow transplantation, leukemia, lymphoma, Hodgkin's disease, multiple myeloma, or generalized malignancy [NOTE: Subjects with prostate or breast cancer who are not on chemotherapeutic drugs (other than hormone blocking drugs), subjects with skin cancer or Kaposi's sarcoma limited to skin who are not receiving radiation therapy or chemotherapy, and subjects with a history of other malignancies who have been disease-free for at least 5 years will be eligible for enrollment.]
* Receipt of any varicella or zoster vaccine prior to study entry
* History of allergy/sensitivity, or hypersensitivity to any vaccine component, including gelatin or neomycin
* Receipt of immunoglobulin or any blood products, other than autologous blood transfusion, given during the 5 months prior to study entry or expected during the 24-week study period
* Receipt of any live virus vaccine within 28 days prior to study entry or during study period
* Receipt of any inactivated vaccine within 7 days prior to study entry or during study period
* Scheduled administration of any live virus vaccine or inactivated vaccine at or between study entry and the Week 12 visit
* Participation in an investigational drug study within the last 30 days prior to study entry
* Use of immunosuppressive therapy. More information can be found in the protocol.
* Any chronic suppressive antiviral therapy with activity against herpes viruses, including but not limited to acyclovir, famciclovir, valacyclovir, ganciclovir, foscarnet, and cidofovir within 7 days prior to study entry or expected use through the 24-week study period except where necessary for acute treatment of intercurrent viral infection.
* Any episode of VZV reactivation in the 12 months prior to study entry
* Active drug or alcohol use, dependence, or any other reason that, in the opinion of the site investigator, would interfere with the study
* Pregnancy (including subjects who are expecting to conceive within 3 months of the second vaccination) or breast feeding
* Any acute intercurrent illness that might interfere with the interpretation of the study
* Significant underlying illness preventing completion of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 395 (Actual)
Dates: Start 2009-04-29 (Actual); Primary Completion 2011-09-22 (Actual); Study Completion 2012-01-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Constance A. Benson, MD, Study Chair — University of California, San Diego; Jeffrey L. Lennox, MD, Study Chair — Emory University
Locations (43):
- United States (43):
  - Alabama Therapeutics CRS, Birmingham, Alabama
  - University of Southern California CRS, Los Angeles, California
  - UCLA CARE Center CRS, Los Angeles, California
  - Stanford CRS, Palo Alto, California
  - Ucsd, Avrc Crs, San Diego, California
  - Ucsf Aids Crs, San Francisco, California
  - Harbor-UCLA Med. Ctr. CRS, Torrance, California
  - University of Colorado Hospital CRS, Aurora, Colorado
  - Denver Public Health CRS, Denver, Colorado
  - Georgetown University CRS (GU CRS), Washington D.C., District of Columbia
  - Univ. of Miami AIDS CRS, Miami, Florida
  - The Ponce de Leon Center CRS, Atlanta, Georgia
  - Northwestern University CRS, Chicago, Illinois
  - Rush Univ. Med. Ctr. ACTG CRS, Chicago, Illinois
  - IHV Baltimore Treatment CRS, Baltimore, Maryland
  - Johns Hopkins Adult AIDS CRS, Baltimore, Maryland
  - Massachusetts General Hospital ACTG CRS, Boston, Massachusetts
  - Brigham and Women's Hosp. ACTG CRS, Boston, Massachusetts
  - Bmc Actg Crs, Boston, Massachusetts
  - Beth Israel Deaconess Med. Ctr., ACTG CRS, Boston, Massachusetts
  - Henry Ford Hosp. CRS, Detroit, Michigan
  - Washington U CRS, St Louis, Missouri
  - Cooper Univ. Hosp. CRS, Camden, New Jersey
  - New Jersey Medical School- Adult Clinical Research Ctr. CRS, Newark, New Jersey
  - Cornell CRS, New York, New York
  - NY Univ. HIV/AIDS CRS, New York, New York
  - HIV Prevention & Treatment CRS, New York, New York
  - Univ. of Rochester ACTG CRS, Rochester, New York
  - Bronx-Lebanon Hosp. Ctr. CRS, The Bronx, New York
  - Chapel Hill CRS, Chapel Hill, North Carolina
  - Duke Univ. Med. Ctr. Adult CRS, Durham, North Carolina
  - Greensboro CRS, Greensboro, North Carolina
  - Univ. of Cincinnati CRS, Cincinnati, Ohio
  - Case CRS, Cleveland, Ohio
  - MetroHealth CRS, Cleveland, Ohio
  - The Ohio State University Medical Center, Columbus, Ohio
  - The Research & Education Group-Portland CRS, Portland, Oregon
  - Hosp. of the Univ. of Pennsylvania CRS, Philadelphia, Pennsylvania
  - Thomas Jefferson Univ. Med. Ctr. CRS, Philadelphia, Pennsylvania
  - Pitt CRS, Pittsburgh, Pennsylvania
  - The Miriam Hosp. ACTG CRS, Providence, Rhode Island
  - Vanderbilt Therapeutics CRS, Nashville, Tennessee
  - University of Washington AIDS CRS, Seattle, Washington

REFERENCES:
- [Background] Gebo KA, Kalyani R, Moore RD, Polydefkis MJ. The incidence of, risk factors for, and sequelae of herpes zoster among HIV patients in the highly active antiretroviral therapy era. J Acquir Immune Defic Syndr. 2005 Oct 1;40(2):169-74. doi: 10.1097/01.qai.0000178408.62675.b0. PMID 16186734
- [Background] Gilderman LI, Lawless JF, Nolen TM, Sterling T, Rutledge RZ, Fernsler DA, Azrolan N, Sutradhar SC, Wang WW, Chan IS, Schlienger K, Schodel F, Silber JL; Zostavax Protocol 010 Study Group. A double-blind, randomized, controlled, multicenter safety and immunogenicity study of a refrigerator-stable formulation of Zostavax. Clin Vaccine Immunol. 2008 Feb;15(2):314-9. doi: 10.1128/CVI.00310-07. Epub 2007 Dec 12. PMID 18077611
- [Background] Holcomb K, Weinberg JM. A novel vaccine (Zostavax) to prevent herpes zoster and postherpetic neuralgia. J Drugs Dermatol. 2006 Oct;5(9):863-6. PMID 17039651
- [Background] Oxman MN, Levin MJ, Johnson GR, Schmader KE, Straus SE, Gelb LD, Arbeit RD, Simberkoff MS, Gershon AA, Davis LE, Weinberg A, Boardman KD, Williams HM, Zhang JH, Peduzzi PN, Beisel CE, Morrison VA, Guatelli JC, Brooks PA, Kauffman CA, Pachucki CT, Neuzil KM, Betts RF, Wright PF, Griffin MR, Brunell P, Soto NE, Marques AR, Keay SK, Goodman RP, Cotton DJ, Gnann JW Jr, Loutit J, Holodniy M, Keitel WA, Crawford GE, Yeh SS, Lobo Z, Toney JF, Greenberg RN, Keller PM, Harbecke R, Hayward AR, Irwin MR, Kyriakides TC, Chan CY, Chan IS, Wang WW, Annunziato PW, Silber JL; Shingles Prevention Study Group. A vaccine to prevent herpes zoster and postherpetic neuralgia in older adults. N Engl J Med. 2005 Jun 2;352(22):2271-84. doi: 10.1056/NEJMoa051016. PMID 15930418
- [Background] Vafai A, Berger M. Zoster in patients infected with HIV: a review. Am J Med Sci. 2001 Jun;321(6):372-80. doi: 10.1097/00000441-200106000-00003. PMID 11417752
- [Derived] Benson CA, Andersen JW, Macatangay BJC, Mailliard RB, Rinaldo CR Jr, Read S, Bozzolo DR, Purdue L, Jennings C, Keefer MC, Glesby M, Tebas P, Russell AF, Martin J, Annunziato P, Popmihajlov Z, Lennox JL. Safety and Immunogenicity of Zoster Vaccine Live in Human Immunodeficiency Virus-Infected Adults With CD4+ Cell Counts >200 Cells/mL Virologically Suppressed on Antiretroviral Therapy. Clin Infect Dis. 2018 Nov 13;67(11):1712-1719. doi: 10.1093/cid/ciy242. PMID 29590326

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first person was accrued on 04/29/2009. Accrual in the high CD4 stratum was closed in 02/2010 (n=203; 152 on ZOSTAVAX and 51 on placebo). Accrual to the low CD4 stratum proceeded more slowly with the last subject enrolled on 06/30/2011 (n=192; 144 on ZOSTAVAX and 48 on placebo). All 43 participating sites enrolled at least 1 subject.
Pre-assignment Details: Enrollment took place in two stages: Stage I were to enroll 48 subjects (24 in the low CD4 stratum and 24 in the high CD4 stratum). Subjects were randomized 3:1 to receive ZOSTAVAX or placebo. Stage II were to enroll approximately 352 subjects who would be randomized and stratified according to the same schedule.
Groups:
- ZOSTAVAX: Participants with CD4 cell counts of 200 cells/uL or greater in Stage 1 and 2, stratified by CD4 cell counts (200-349 cells/uL vs. >=350 cells/uL), will be given one dose of ZOSTAVAX (Zoster Vaccine Live) at Day 0 and Week 6 and will be followed for at least 42 days after each vaccination after which a safety assessment will be conducted.
- Placebo: Participants with CD4 cell counts of 200 cells/uL or greater in Stage 1 and 2, stratified by CD4 cell counts (200-<349 cells/uL vs. >=350 cells/uL), will be given one dose of placebo at Day 0 and Week 6 and will be followed for at least 42 days after each vaccination afer which a safety assessment will be conducted
Period: Overall Study
Arm/Group | ZOSTAVAX | Placebo
Started | 296 (One subject cannot adhere to protocol requirement and was off study with no vaccine.) | 99 (Two subjects (one found ineligible and one withdrew consent) were off study with no vaccine.)
Completed | 291 | 97
Not Completed | 5 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Incarceration | 1 | 0
Not completed — Site Closure | 1 | 0
Not completed — Cannot Adhere to Protocol Requirement | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ZOSTAVAX | Placebo | Total
Number analyzed (Participants) | 296 | 99 | 395
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 285 | 94 | 379
  >=65 years | 11 | 5 | 16
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 49 [44 to 56] | 49 [44 to 55] | 49 [44 to 56]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 18 | 62
  Male | 252 | 81 | 333
Race/Ethnicity, Customized [Number; unit: participants]
  White Non-Hispanic | 141 | 44 | 185
  Black Non-Hispanic | 90 | 26 | 116
  Hispanic (regardless of race) | 60 | 27 | 87
  Asian, Pacific islander | 1 | 1 | 2
  American Indian, Alaskan Native | 2 | 1 | 3
  More than one race | 1 | 0 | 1
  Unknown/missing | 1 | 0 | 1
IV drug history [Number; unit: participants]
  Never | 244 | 86 | 330
  Previously | 52 | 13 | 65
Nadir CD4 [Median (Inter-Quartile Range); unit: cells/µL] | 197 [109 to 287] | 178 [104.5 to 285] | 188 [108 to 287]
Screen CD4 [Median (Inter-Quartile Range); unit: cells/µL] | 373 [286 to 634.5] | 353 [278 to 561] | 372 [286 to 606]
Entry CD4 [Median (Inter-Quartile Range); unit: cells/µL] | 399 [282 to 607] | 362 [276 to 579] | 394 [281 to 605]
HIV-1 RNA [Median (Inter-Quartile Range); unit: log10 copies/mL] | 1.68 [1.68 to 1.70] | 1.68 [1.68 to 1.70] | 1.68 [1.68 to 1.70]
Prior History of AIDS [Number; unit: participants]
  Yes | 288 | 97 | 385
  No | 8 | 2 | 10
History of Chickenpox [Number; unit: participants]
  >5 years | 219 | 77 | 296
  Zoster/no Chickpox | 17 | 7 | 24
  None | 60 | 15 | 75
History of most recent Zoster [Number; unit: participants]
  0-1 year | 2 | 1 | 3
  >1-2 years | 13 | 1 | 14
  >2-5 years | 23 | 7 | 30
  >5 years | 65 | 22 | 87
  None | 193 | 68 | 261
Duration from Historary Retinal Necrosis [Number; unit: participants]
  >5 years | 2 | 0 | 2
  None | 294 | 99 | 393

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Composite Safety Endpoint of the Occurrence of Serious Adverse Events (SAEs) or Division of AIDS (DAIDS) Grade 3 and 4 Signs and Symptoms, Excluding SAEs Related to Trauma
Description: Although the study was designed as a randomized trial, it was not powered to detect safety related differences between treatment arms. The safety of ZOSTAVAX was determined by comparing the number of subjects from the active arm who experienced safety endpoint to the number from a pre-specified decision rule, which was calculated based on a similar population and calibrated using the number of safety endpoints observed from the placebo arm. The pre-specified decision rule is that ZOSTAVAX would be considered to have acceptable safety if no more than 18 subjects experience a study-defined composite safety endpoint.
Time Frame: During the 6 week study period after receipt of any dose of ZOSTAVAX
Population: Subjects who received at least one dose of study vaccine/placebo
Measure: Number; unit: participants
Arm/Group | ZOSTAVAX | Placebo
Number analyzed (Participants) | 295 | 97
participants | 15 [0.029 to 0.082] | 2 [0.003 to 0.073]

2. Secondary Outcome: VZV Antibodies as Measured by gpELISA
Description: VZV antibody titer measured by gpELISA after one or two doses of ZOSTAVAX/placebo
Time Frame: Within 6 weeks following one or two doses of ZOSTAVAX
Population: Subjects with both baseline gpELISA result and at least one post vaccination gpELISA result available
Measure: Mean (Standard Deviation); unit: log gpELISA antibody titer
Arm/Group | ZOSTAVAX | Placebo
Number analyzed (Participants) | 280 | 96
log gpELISA antibody titer
  Baseline | 5.68 (1.03) | 5.52 (1.26)
  6 weeks after 1st ZOSTAVAX/Placebo | 6.28 (0.92) | 5.57 (1.27)
  6 weeks after 2nd ZOSTAVAX/Placebo | 6.27 (0.87) | 5.52 (1.27)
Statistical Analysis 1: Comparison: ZOSTAVAX vs Placebo; Null hypothesis: VZV antibody titer measured by gpELISA, after 1 or 2 doses of ZOSTAVAX/placebo is the same between ZOSTAVAX arm and the placebo arm; Test type: Superiority or Other; p < .001, Linear mixed effect model — The p-value was adjusted for baseline gpELISA titer, measurement time (week 6 vs. week 12), CD4 stratum and age; Natural log transformed gpELISA titers after one or two doses of vaccine was modeled; Mean Difference (Final Values) = 0.57, 95% CI 2-sided [0.45 to 0.69], Standard Error of Mean 0.06

3. Secondary Outcome: Geometric Mean Fold Rise (GMFR) in VZV ELISpot Responses
Description: VZV-specific cellular immune responses in peripheral blood mononuclear cells (PBMC) were tested by ELISpot assay in a subset of participants pooled across CD4 strata. GMFR is the geometric mean of the ratios of Week 6 or Week 12 post-vaccination antibody to the pre-vaccination antibody.
Time Frame: Entry, Week 6, Week 12
Population: Number of participants with ELISpot results available at entry and at the post-entry week (week 6 or week 12, respectively).
Measure: Geometric Mean (90% Confidence Interval); unit: fold rise
Arm/Group | ZOSTAVAX | Placebo
Number analyzed (Participants) | 56 | 18
fold rise
  Week 6 GMFR | 1.8 [0.8 to 3.7] | 0.4 [0.2 to 1.1]
  Week 12 GMFR: number analyzed (Participants) | 54 | 16
  Week 12 GMFR | 3.8 [1.8 to 8.0] | 1.1 [0.3 to 3.4]

ADVERSE EVENTS:
Time Frame: From study entry to study exit, approximately 24 weeks.
Arm/Group | ZOSTAVAX | Placebo
All-Cause Mortality (participants affected / at risk) | 1/296 | 0/99
Serious Adverse Events (participants affected / at risk) | 15/296 | 7/99
Other Adverse Events (participants affected / at risk) | 98/296 | 15/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ZOSTAVAX (N=296) | Placebo (N=99)
Atrial fibrillation (Cardiac disorders) | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Gun shot wound (Injury, poisoning and procedural complications) | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung carcinoma cell type unspecified recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Migraine (Nervous system disorders) | 1 | 0
Bulimia nervosa (Psychiatric disorders) | 1 | 0
Delirium (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ZOSTAVAX (N=296) | Placebo (N=99)
Injection site erythema (General disorders) | 34 | 0
Injection site pain (General disorders) | 52 | 4
Injection site swelling (General disorders) | 16 | 0
Pyrexia (General disorders) | 13 | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 17 | 1
Headache (Nervous system disorders) | 18 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with the Clinical Trials Agreement between NIAID (DAIDS) and company collaborators, NIAID (DAIDS) provides companies with a copy of any abstract, press release, or manuscript prior to submission for publication with sufficient time for company review and comment. The publication/other disclosure can be delayed for up to 30 additional business days for manuscripts and five (5) business days for abstracts, to preserve U.S. or foreign patent or other intellectual property rights.